CLINICAL TRIAL: NCT05196256
Title: A Double-blind, Randomized, Controlled, Pilot Study Comparing Three Different Anesthesic Techniques for Pregnant Women in Labour: Dural Puncture Epidural, Epidural and Combined Spinal Epidural. Evaluation of the Pain Control and the Hypotension Incidence All Along the Labour and Delivery
Brief Title: Study Comparing Dural Puncture Epidural With Epidural and Combined Spinal Epidural Anesthesia for Obstetric Analgesia.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head, department of Anesthesiology, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUB-MAT-DPE
Record Dates: First submitted 2021-12-30; First posted 2022-01-19 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Obstetric Pain; Analgesia
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Analgesia, Epidural; Sufentanil; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized by envelopes. A non-blinded anesthesiologists will perform the anesthetics technique and leave the room immediately; a blinded anesthesiologists will do the data collection and act according to protocol if the patient in case of pain non controllable by the patient controlled anesthesia, in case of hypotension or any other possible complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dural Puncture Epidural group (DPE) (Experimental): Dural puncture with a 25 Gauge needle, then placement of the epidural catheter (Tuohy 18 Gauge). The medication consists of Levobupivacaine 0.0625% and Sufentanyl 0.25 mcg/mL, both administered epidurally with a programmed intermittent bolus mode (PIB) and patient controlled epidural analgesia (PCEA). An initial fractionated bolus of 20 mL will be administered epidurally, then automatic intermittent bolus of 10 mL will be administered, the first one after 30 min and then every 40min. PCEA pump will allow 10 mL every 20 min, all along the dilatation and expulsion period.
  Interventions: Procedure: Dural puncture; Drug: Sufentanyl/Levobupivacaine
- Epidural group (EP) (Active Comparator): Placement of an epidural catheter through a 18 Gauge Tuohy needle. The medication consists of Levobupivacaine 0.0625% and Sufentanyl 0.25 mcg/mL, both administered epidurally with a programmed intermittent boluses mode (PIB) and patient controlled epidural analgesia (PCEA); An initial fraction bolus of 20ml will be administered epidurally, then automatic intermittent bolus of 10 mL will be administered, the first one after 30 min and then every 40 min. PCEA pump will allow 10 mL every 20 min, all along the dilatation and expulsion period.
  Interventions: Procedure: Epidural analgesia; Drug: Sufentanyl/Levobupivacaine
- Combined Spinal-Epidural group (CSE) (Active Comparator): Spinal injection through a 25 Gauge needle of Levobupivacaine 2.5mg and Sufentanyl 2.5 mcg in a total volume of 2 mL, placing an epidural catheter through a Tuohy 18 Gauge needle. The epidural medication consists of Levobupivacaine 0.0625% and Sufentanyl 0.25 mcg/mL. The epidural medication is administered on a programmed intermittent bolus mode (PIB) and patient controlled epidural analgesia (PCEA). An initial fractioned bolus of 20 mL will be administered epidurally 30 min after the intrathecal injection, then automatic intermittent bolus of 10 mL will be administered, the first one after 30 min and then every 40 min. PCEA pump will allow 10 mL every 20min, all along the dilatation and expulsion period.
  Interventions: Procedure: Combined spinal epidural analgesia; Drug: Sufentanyl/Levobupivacaine

INTERVENTIONS:
Procedure: Dural puncture — Dural puncture with a 25 Gauge needle without injection of local anesthetics into the dural space
  Arms: Dural Puncture Epidural group (DPE)
Procedure: Combined spinal epidural analgesia — Standard epidural preceded by a dural puncture with a 25G sequential needle and intrathecal injection of 2.5 ug of Sufentanil and 2.5 mg of normobaric Levobupivacaine
  Arms: Combined Spinal-Epidural group (CSE)
Procedure: Epidural analgesia — Epidural analgesia
  Arms: Epidural group (EP)
Drug: Sufentanyl/Levobupivacaine — Epidural analgesia

SUMMARY:
This will be a prospective, randomized, double blind, controlled clinical trial.

Epidural analgesia (EP) is currently the method of choice to ensure the comfort of the parturient during childbirth. Technical and pharmacological advances in recent years have made it possible to provide patients with high quality analgesia with individualized control, associated with extremely limited motor block. However, sometimes this technique fails due to a prolonged delay in action, or insufficient sensory block.

An alternative technique has become popular in recent years, the combined peri-spinal anesthesia also called sequential (CSE). It combines the administration of low doses of local anesthetics and/or intrathecal opiates before the placement of the catheter in the epidural space and the use of the catheter as in a classical technique. This technique would allow a more rapid onset of analgesia, a more complete relief of the patient, and a lower degree of failure. However, it could be accompanied by a greater risk of maternal hemodynamic instability, fetal bradycardia, and a longer expulsion period. In addition, the effectiveness of the catheter injection can only be assessed when the effects of the spinal injected drugs have worn off.

In order to limit these undesirable effects, it has been proposed to perform a dural puncture as performed in the sequential technique but without intrathecal drug injection (DPE). In this way, a "tunnel" is created, allowing the diffusion of drugs from the epidural space to the subarachnoid space. Thus, the initiation of anesthesia would be faster with a lower risk of lateralization compared to the standard epidural, also allowing a decrease in the consumption of local anesthetics and without the undesirable effects of the sequential. Although this technique recently introduced in obstetrical analgesia appears promising, very few studies to date have evaluated its effectiveness and safety.

The hypothesis of the study is that the Epidural with Dural puncture (DPE) provides a higher quality of analgesia than standard epidural while having fewer adverse effects than combined epidural, in particular a lower incidence of maternal hypotension.

The primary objectives are:

* testing the quality of analgesia with DPE compared to PE and CSE. This will be assessed by determining the area under the curve of Visual Analog Scale (VAS) measurements observed from the beginning of obstetric analgesia and throughout the delivery.
* testing the rate of maternal hypotension with DPE compared with PE and CSE, with hypotension defined as a decrease in systolic blood pressure (SBP) greater than 15% from the SBP measured at the time of the parturient arrival in the labor room, a SBP < 90 mmHg, or any decrease in pressure associated with disabling symptomatology (dizziness, yawning, nausea).

For this purpose, the investigators will randomize a total of 90 patients, 30 in each of the groups. The patients will receive one of the three techniques, all of them will benefit from the administration of epidural analgesia with low concentration local anesthetics and opioids on a Intermittent bolus modus (PIB). Patients assigned to the combined spinal epidural modus will receive a injection of a small quantity of local anesthetics and opioids (Levobupivacaine 2.5mg and Sufentanyl 2.5 mcg) in the intrathecal space. A non-blinded anesthesiologists will perform the anesthetics technique and leave the room immediately; a blinded anesthesiologists will do the data collection and act according to protocol if the patient in case of pain non controllable by the patient controlled anesthesia, in case of hypotension or any other possible complications.

Data collection will take place before starting the locoregional anesthesia technique, at the moment when the anesthetists non blinded leaves the room, 10 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours after the start of the analgesia and at the moment of the expulsion of the baby.

Patients and care providers will be blinded to which technic is being given. Data will be statistically analyzed using area under the curve and two-dimension variance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term (37-42 weeks of amenorrhea)
* American Society of Anesthesiologists (ASA) class 1 or 2
* no language barrier, i.e; speaking French, Dutch or English or accompanied by a reliable translator
* single pregnancy
* Parity 1 , 2 or 3
* cephalic fetal presentation
* active labor with cervical dilatation less than 5 cm

Exclusion Criteria:

* Contraindications to neuraxial anesthesia
* major pathologies of pregnancy (preeclampsia)
* decompensated gestational diabetes
* diabetes type 1 or 2
* known serious fetal pathology
* maternal previous diseases increasing the risk of caesarean section (caesarean section, uterine malformation, scarred uterus, surgery of the uterine cervix)
* fourth or more deliveries
* extreme pre-pregnancy BMI (< 18 or > 40)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of the pain visual analog scale (VAS) | 10 minutes after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 15 minutes after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 30 minutes after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 1 hour after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 2 hours after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 3 hours after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 4 hours after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | 6 hours after the start of the anesthesia technique
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Area under the curve of the pain visual analog scale (VAS) | From the start of the anesthesia technique until delivery of the baby (max up to 24 hours)
  Evaluation of the quality of analgesia, calculated from the area under the curve of the VAS. The measurements will be performed by a "blind" team member.
Incidence of maternal hypotension | 24 hours
  To test whether DPE is accompanied by a lower incidence of maternal hypotension than CSE. For the purposes of this study, hypotension is defined as a decrease of more than 15% in systolic blood pressure (SBP) from the first pressure taken when the patient was admitted to the labor room, SBP < 90 mm Hg, or any decrease in SBP accompanied by symptomatology (malaise, nausea) requiring rescue treatment. Incidence will be measured as percentage of patients presenting a hypotension according to this definition.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sodha S, Reeve A, Fernando R. Central neuraxial analgesia for labor: an update of the literature. Pain Manag. 2017 Sep;7(5):419-426. doi: 10.2217/pmt-2017-0010. Epub 2017 Sep 22. PMID 28936908
- [Background] Sng BL, Kwok SC, Sia AT. Modern neuraxial labour analgesia. Curr Opin Anaesthesiol. 2015 Jun;28(3):285-9. doi: 10.1097/ACO.0000000000000183. PMID 25827278
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Pan PH, Bogard TD, Owen MD. Incidence and characteristics of failures in obstetric neuraxial analgesia and anesthesia: a retrospective analysis of 19,259 deliveries. Int J Obstet Anesth. 2004 Oct;13(4):227-33. doi: 10.1016/j.ijoa.2004.04.008. PMID 15477051
- [Background] Bucstain C, Garmi G, Zafran N, Zuarez-Easton S, Carmeli J, Salim R. Risk factors and peripartum outcomes of failed epidural: a prospective cohort study. Arch Gynecol Obstet. 2017 May;295(5):1119-1125. doi: 10.1007/s00404-017-4337-5. Epub 2017 Mar 10. PMID 28283828
- [Background] Gambling D, Berkowitz J, Farrell TR, Pue A, Shay D. A randomized controlled comparison of epidural analgesia and combined spinal-epidural analgesia in a private practice setting: pain scores during first and second stages of labor and at delivery. Anesth Analg. 2013 Mar;116(3):636-43. doi: 10.1213/ANE.0b013e31827e4e29. Epub 2013 Feb 11. PMID 23400985
- [Background] Goodman SR, Smiley RM, Negron MA, Freedman PA, Landau R. A randomized trial of breakthrough pain during combined spinal-epidural versus epidural labor analgesia in parous women. Anesth Analg. 2009 Jan;108(1):246-51. doi: 10.1213/ane.0b013e31818f896f. PMID 19095858
- [Background] Booth JM, Pan JC, Ross VH, Russell GB, Harris LC, Pan PH. Combined Spinal Epidural Technique for Labor Analgesia Does Not Delay Recognition of Epidural Catheter Failures: A Single-center Retrospective Cohort Survival Analysis. Anesthesiology. 2016 Sep;125(3):516-24. doi: 10.1097/ALN.0000000000001222. PMID 27380107
- [Background] Heesen M, Van de Velde M, Klohr S, Lehberger J, Rossaint R, Straube S. Meta-analysis of the success of block following combined spinal-epidural vs epidural analgesia during labour. Anaesthesia. 2014 Jan;69(1):64-71. doi: 10.1111/anae.12456. Epub 2013 Oct 28. PMID 24164577
- [Background] Hattler J, Klimek M, Rossaint R, Heesen M. The Effect of Combined Spinal-Epidural Versus Epidural Analgesia in Laboring Women on Nonreassuring Fetal Heart Rate Tracings: Systematic Review and Meta-analysis. Anesth Analg. 2016 Oct;123(4):955-64. doi: 10.1213/ANE.0000000000001412. PMID 27509225
- [Background] Simmons SW, Taghizadeh N, Dennis AT, Hughes D, Cyna AM. Combined spinal-epidural versus epidural analgesia in labour. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003401. doi: 10.1002/14651858.CD003401.pub3. PMID 23076897
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Background] Poma S, Scudeller L, Verga C, Mirabile G, Gardella B, Broglia F, Ciceri M, Fuardo M, Pellicori S, Gerletti M, Zizzi S, Masserini E, Delmonte MP, Iotti GA. Effects of combined spinal-epidural analgesia on first stage of labor: a cohort study. J Matern Fetal Neonatal Med. 2019 Nov;32(21):3559-3565. doi: 10.1080/14767058.2018.1467892. Epub 2018 May 17. PMID 29768964
- [Background] Van de Velde M, Teunkens A, Hanssens M, Vandermeersch E, Verhaeghe J. Intrathecal sufentanil and fetal heart rate abnormalities: a double-blind, double placebo-controlled trial comparing two forms of combined spinal epidural analgesia with epidural analgesia in labor. Anesth Analg. 2004 Apr;98(4):1153-1159. doi: 10.1213/01.ANE.0000101980.34587.66. PMID 15041616
- [Background] Cappiello E, O'Rourke N, Segal S, Tsen LC. A randomized trial of dural puncture epidural technique compared with the standard epidural technique for labor analgesia. Anesth Analg. 2008 Nov;107(5):1646-51. doi: 10.1213/ane.0b013e318184ec14. PMID 18931227
- [Background] Wilson SH, Wolf BJ, Bingham K, Scotland QS, Fox JM, Woltz EM, Hebbar L. Labor Analgesia Onset With Dural Puncture Epidural Versus Traditional Epidural Using a 26-Gauge Whitacre Needle and 0.125% Bupivacaine Bolus: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):545-551. doi: 10.1213/ANE.0000000000002129. PMID 28622178
- [Background] Heesen M, Rijs K, Rossaint R, Klimek M. Dural puncture epidural versus conventional epidural block for labor analgesia: a systematic review of randomized controlled trials. Int J Obstet Anesth. 2019 Nov;40:24-31. doi: 10.1016/j.ijoa.2019.05.007. Epub 2019 May 13. PMID 31281033
- [Background] Layera S, Bravo D, Aliste J, Tran DQ. A systematic review of DURAL puncture epidural analgesia for labor. J Clin Anesth. 2019 Mar;53:5-10. doi: 10.1016/j.jclinane.2018.09.030. Epub 2018 Sep 28. PMID 30273698
- [Background] Thomas JA, Pan PH, Harris LC, Owen MD, D'Angelo R. Dural puncture with a 27-gauge Whitacre needle as part of a combined spinal-epidural technique does not improve labor epidural catheter function. Anesthesiology. 2005 Nov;103(5):1046-51. doi: 10.1097/00000542-200511000-00019. PMID 16249679
- [Background] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Background] Song Y, Du W, Zhou S, Zhou Y, Yu Y, Xu Z, Liu Z. Effect of Dural Puncture Epidural Technique Combined With Programmed Intermittent Epidural Bolus on Labor Analgesia Onset and Maintenance: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):971-978. doi: 10.1213/ANE.0000000000004768. PMID 32282386
- [Background] Abrao KC, Francisco RPV, Miyadahira S, Cicarelli DD, Zugaib M. Elevation of uterine basal tone and fetal heart rate abnormalities after labor analgesia: a randomized controlled trial. Obstet Gynecol. 2009 Jan;113(1):41-47. doi: 10.1097/AOG.0b013e31818f5eb6. PMID 19104358
- [Background] Everaert N, Coppens M, Vlerick P, Braems G, Wouters P, De Hert S. Combined spinal epidural analgesia for labor using sufentanil epidurally versus intrathecally: a retrospective study on the influence on fetal heart trace. J Perinat Med. 2015 Jul;43(4):481-4. doi: 10.1515/jpm-2014-0077. PMID 24922321